CLINICAL TRIAL: NCT04750902
Title: A Phase 2 Randomized, Double-blind, Active-controlled Multi-center Clinical Trial to Assess the Safety and the Anti-caries Efficacy of COL 101 (Arginine) Non-fluoride Dentifrices With 1.5%, 4.0% and 8.0% Arginine Each in Comparison With 0.24% Sodium Fluoride (1100 Ppm F) Dentifrice Control in 10 to 14-year-old Children
Brief Title: A Clinical Trial to Assess the Safety and the Anti-caries Efficacy of COL 101 (Arginine) Non-fluoride Dentifrices in Comparison With 0.24% Sodium Fluoride (1100 Ppm F) Dentifrice Control in 10 to 14-year-old Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CRO-2020-CAR-ARG-ED
Record Dates: First submitted 2021-02-08; First posted 2021-02-11 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Dental Caries
Keywords: fluoride; arginine; prevention; caries; ICDAS; DMFS
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 0.24% Sodium Fluoride Dentifrice (Active Comparator): Toothpaste
  Interventions: Drug: 0.24% Sodium Fluoride Dentifrice
- 1.5% Arginine Dentifrice (Experimental): Toothpaste
  Interventions: Drug: 1.5% Arginine Dentifrice
- 4.0% Arginine Dentifrice (Experimental): Toothpaste
  Interventions: Drug: 4.0% Arginine Dentifrice
- 8.0% Arginine Dentifrice (Experimental): Toothpaste
  Interventions: Drug: 8.0% Arginine Dentifrice

INTERVENTIONS:
Drug: 0.24% Sodium Fluoride Dentifrice — Whole mouth brushing with a toothpaste, 2 times/day for 2 minutes each time for the duration of the study
  Arms: 0.24% Sodium Fluoride Dentifrice
Drug: 1.5% Arginine Dentifrice — Whole mouth brushing with a toothpaste, 2 times/day for 2 minutes each time for the duration of the study
  Arms: 1.5% Arginine Dentifrice
Drug: 4.0% Arginine Dentifrice — Whole mouth brushing with a toothpaste, 2 times/day for 2 minutes each time for the duration of the study
  Arms: 4.0% Arginine Dentifrice
Drug: 8.0% Arginine Dentifrice — Whole mouth brushing with a toothpaste, 2 times/day for 2 minutes each time for the duration of the study
  Arms: 8.0% Arginine Dentifrice

SUMMARY:
The objective of this study is to assess the safety and to evaluate the anti-caries efficacy of COL101 (arginine) non-fluoride dentifrices compared to a 0.24% sodium fluoride dentifrice in 10-14 year-old children over a one year period.

ELIGIBILITY:
Inclusion Criteria:

* Subjects meeting all criteria below will be included in the study:

  1. Subject assent and parental/guardian informed consent for voluntary participation.
  2. Willingness and ability to use the assigned products according to instructions, availability for all appointments and likelihood of completing the clinical trial.
  3. Children ages 10-14 years at baseline.
  4. Presence of permanent second molars or evidence of at least one permanent second molar erupting as indicated by cuspal break through the mucosa.
  5. Good general health as evidenced by a review of the medical history.
  6. Subjects who, at study entry, have present two or more active caries lesions (ICDAS scores of 2 or greater) in permanent teeth and previous caries experience (DMFT >1), D= Decayed is defined as ICDAS scores of 3 or greater

Exclusion Criteria:

* Subjects presenting any of the criteria below will be excluded from the study:

  1. Presence of fixed or removable prosthetic appliance or orthodontic treatment involving more than four permanent teeth.
  2. Use of medication that could increase the risk of developing dental caries, i.e.

     medications that reduce saliva flow and those with high sugar content.
  3. Long-term antibiotic therapy.
  4. Children with a confirmed diagnosis of cognitive and/or motor impairment.
  5. Severe malocclusion.
  6. Subjects who, at study entry, have present severe caries (ICDAS 5 or 6) on five or more permanent teeth.
  7. Evidence of moderate to severe periodontal disease.
  8. Participation in any other clinical study within the 30 days preceding the start of the clinical study.
  9. Known history of allergies or other adverse reactions to arginine, or oral care products, or their ingredients.
  10. Self-reported history of being currently pregnant, intending to become pregnant during the trial period or breast-feeding.

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2000 (Actual)
Dates: Start 2021-01-21 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint will be the incremental subject-wise Decayed Missing Filled Surfaces (DMFS) score after one year of product use | one year
  the minimum score is 0, maximum score is 4/5 depending on the tooth number and a higher score represents a worse outcome

SECONDARY OUTCOMES:
Incremental subject-wise Decayed Missing Filled Surfaces (DFMS) score after 6-months of product use; | after 6 months
  the minimum score is 0, maximum score is 4/5 depending on the tooth number and a higher score represents a worse outcome
Incremental subject-wise Decayed Missing Filled Surfaces (DFMS) score between 6- months and one year of product use. | between 6-months and one year
  the minimum score is 0, maximum score is 4/5 depending on the tooth number and a higher score represents a worse outcome
Clinically significant change in International Caries Detection and Assessment System (ICDAS) severity scores between the baseline and the six-month and one-year examinations and between the six-month and one-year examinations. | between 6-months and one year
  the minimum score is 0, maximum score is 6 and a higher score represents a worse outcome
Clinically significant changes indicating caries progression are changes in ICDAS severity values from 0 to 2 or higher, from 1 or 2 to 3 or higher, or from 3 or 4 to 5 or 6. | 6 months
Clinically significant changes indicating caries regression are changes in ICDAS severity values from 2 or higher to 0 or 1. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Maria E Ryan, DDS PhD, Study Director — Colgate-Palmolive Company
Locations (9):
- United States (8):
  - Loma Linda University School of Dentistry, Loma Linda, California
  - University of Florida College of Dentistry, Gainesville, Florida
  - Indiana University School of Dentistry, Indianapolis, Indiana
  - Tufts University School of Dental Medicine, Boston, Massachusetts
  - The Forsyth Institute, Boston, Massachusetts
  - University at Buffalo School of Dental Medicine, Buffalo, New York
  - University of Pennsylvania School of Dental Medicine, Philadelphia, Pennsylvania
  - UT Health San Antonio School of Dentistry, San Antonio, Texas
- University of Puerto Rico School of Dental Medicine, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No